CLINICAL TRIAL: NCT03382509
Title: A Phase I, Open-label, Single and Multiple Dose Trial to Investigate Metabolism and Pharmacokinetics of [14C]BI 1467335 Administered as Oral Solution in Healthy Male Volunteers
Brief Title: This Study Tests BI 1467335 in Healthy Male Volunteers. The Study Tests How Different Doses of BI 1467335 Are Taken up and Handled by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1386-0011; 2017-002879-26 (EudraCT Number)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Dose Group (Experimental)
  Interventions: Drug: [14C]BI 1467335
- Multiple Dose Group (Experimental)
  Interventions: Drug: BI 1467335

INTERVENTIONS:
Drug: [14C]BI 1467335 — Once Daily
  Arms: Single Dose Group
Drug: BI 1467335 — Twice Daily
  Arms: Multiple Dose Group

SUMMARY:
Primary objective mass balance, excretion pathways and metabolism following a single oral dose of [14C]BI 1467335 given to healthy male subjects (a selected number of subjects will be treated with [14C]BI 1467335 after a preceding 27 days treatment with non-radiolabelled compound of BI 1467335 QD).

Secondary objectives is to investigate the basic pharmacokinetics after single and multiple doses of BI 1467335 and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram, and clinical laboratory tests
* Age of 30 to 65 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Subjects who are sexually active must use, with their partner, highly effective contraception from the time of administration of trial medication until 4 months after administration of trial medication. --Adequate methods are:

  * Condoms plus use of hormonal contraception by the female partner that started at least 2 months prior to administration of trial medication (e.g., implants, injectables, combined oral or vaginal contraceptives, intrauterine device) or
  * Condoms plus surgical sterilization (vasectomy at least 1 year prior to enrolment) or
  * Condoms plus surgically sterilised partner (including hysterectomy) or
  * Condoms plus intrauterine device or
  * Condoms plus partner of non-childbearing potential (including homosexual men)

    * Subjects are required to use condoms to prevent unintended exposure of the partner to the study drug via seminal fluid.
    * Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, with their partner, they must comply with the contraceptive requirements detailed above

Exclusion Criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram) is deviating from normal and judged as clinically relevant by the investigator
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Clinically significant gastrointestinal, hepatic, renal, respiratory (including but not limited to interstitial lung disease), cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Within 30 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 5 cigarettes or 1 cigar or 1 pipe per day)
* Inability to refrain from smoking on specified trial days
* Average intake of more than 24 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTcF intervals that are repeatedly greater than 450 ms) or any other relevant Electrocardiogram finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences Onderzoekscentrum Martini, Groningen, Netherlands

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, phase I, single-arm, and 2 study parts trial with either single or multiple dose in healthy male participants. The single dose (SD) and multiple dose (MD) parts of the trial were conducted in different participants. The trial started with the MD part, while the SD part was scheduled close to Day 28 of the MD part.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensured that all participants met all inclusion/exclusion criteria. Participants were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Groups:
- BI 1467335 10 Milligram (mg) (SD): Participants were administered single dose of 10 milligram (mg) carbon 14 (14C) labelled BI 1467335 solution orally on Day 1 with 240 milliliter (mL) of water after an overnight fast of at least 10 hours.
- BI 1467335 10 mg (MD): Participants were administered once daily 10 mg (2*5 mg) BI 1467335 non-radiolabelled film-coated tablets Day 1 to Day 27 and Day 29 to a maximum of Day 40 orally with 240 milliliter (mL) of water. On Day 28 a single dose of 14C BI 1467335 oral solution was administered.
Period: Overall Study
Arm/Group | BI 1467335 10 Milligram (mg) (SD) | BI 1467335 10 mg (MD)
Started (Started are treated) | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This set included all participants who received at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1467335 10 Milligram (mg) (SD) | BI 1467335 10 mg (MD) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (4.5) | 57.3 (10.9) | 58.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Fraction of [14C]-Radioactivity Excreted in Urine as Percentage of the Administered Oral Dose Over the Time Interval From 0 to the Last Quantifiable Time Point (fe(Urine,0-t2))
Description: fe(urine, 0-t2), fraction of [14C]-radioactivity excreted in urine as percentage of the administered oral dose over the time interval from 0 to the last quantifiable time point.
Time Frame: 2 hours (h) prior to drug intake at Day 1 (SD group) and at the following intervals on Day 1 (SD group) and Day 28 (MD group): 0 to 4, 4 to 8, 8 to 12, 12 to 24 hours and every 24 hours thereafter from day 1 to day 14 following drug intake.
Population: Pharmacokinetic parameter analysis set (PKS): This subject set included all subjects of the TS who provided at least 1 primary or secondary PK parameter that was not excluded because of protocol deviations relevant to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose excreted
Arm/Group | BI 1467335 10 Milligram (mg) (SD) | BI 1467335 10 mg (MD)
Number analyzed (Participants) | 8 | 8
Percentage of dose excreted | 79.0 (2.68) | 83.7 (2.12)

2. Primary Outcome: Fraction of [14C]-Radioactivity Excreted in Faeces as Percentage of the Administered Oral Dose Over the Time Interval From 0 to the Last Quantifiable Time Point (fe(Faeces,0-t2))
Description: fe(faeces,0-t2), fraction of [14C]-radioactivity excreted in faeces as percentage of the administered oral dose over the time interval from 0 to the last quantifiable time point.
  Time frame: 648 to 672 h, 672 to 696, 696 to 720, 720 to 744, 744to 768, 768 to 792, 792 to 816, 816 to 840, 840 to 864, 864 to 888, 888 to 912, 912 to 936, 936 to 960, 960 to 984, and 984 to 1008 after the dispense of study medication at Day 1 for the MD group.
Time Frame: 2 hours (h) prior to drug intake at Day 1 (SD group) and at the following intervals on Day 1 (SD group) and Day 28 (MD group): every 24 hours from day 1 to day 14 following drug intake.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose excreted
Arm/Group | BI 1467335 10 Milligram (mg) (SD) | BI 1467335 10 mg (MD)
Number analyzed (Participants) | 8 | 8
Percentage of dose excreted | 12.6 (15.1) | 8.82 (13.9)

3. Secondary Outcome: Maximum Measured Concentration of 14C-BI 1467335-Equivalence (EQ) in Plasma After Single Oral Administration of [14C]BI 1467335 (Cmax)
Description: Cmax, maximum measured concentration of 14C-BI 1467335-Equivalence (EQ) in plasma after single oral administration of [14C]BI 1467335 is presented.
Time Frame: Pharmacokinetic samples were collected at 2 hours (h) prior to drug administration and at 0.33, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 192, 240, 288, 336, 485, 653, 821, 989 and 1157 h after drug administration on Day 1.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/ Liter (nmol/L)
Arm/Group | BI 1467335 10 Milligram (mg) (SD)
Number analyzed (Participants) | 8
nanomole/ Liter (nmol/L) | 503.0 (12.7)

4. Secondary Outcome: Area Under the Concentration-time Curve of 14C-BI 1467335-Equivalence (EQ) Over the Time Interval From 0 to the Last Quantifiable Time Point in Plasma After Single Oral Administration of [14C]BI 1467335 (AUC0-tz)
Description: AUC0-tz, area under the concentration-time curve of 14C-BI 1467335-Equivalence(EQ) over the time interval from 0 to the last quantifiable time point in plasma after single oral administration of [14C]BI 1467335 is presented.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole * hour/Liter (nmol*h/L)
Arm/Group | BI 1467335 10 Milligram (mg) (SD)
Number analyzed (Participants) | 8
nanomole * hour/Liter (nmol*h/L) | 72900.0 (18.1)

5. Secondary Outcome: Maximum Measured Concentration of BI 1467335 in Plasma After Single Oral Administration of [14C]BI 1467335 (Cmax)
Description: Cmax, maximum measured concentration of BI 1467335 in plasma after single oral administration of [14C]BI 1467335 is presented.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1467335 10 Milligram (mg) (SD)
Number analyzed (Participants) | 8
nanomole/Liter (nmol/L) | 2.88 (146.00)

6. Secondary Outcome: Area Under the Concentration-time Curve of BI 1467335 Over the Time Interval From 0 to the Last Quantifiable Time Point in Plasma After Single Oral Administration of [14C]BI 1467335 (AUC0-tz)
Description: AUC0-tz, area under the concentration-time curve of BI 1467335 over the time interval from 0 to the last quantifiable time point in plasma after single oral administration of [14C]BI 1467335 is presented.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole * hour/Liter (nmol*h/L)
Arm/Group | BI 1467335 10 Milligram (mg) (SD)
Number analyzed (Participants) | 8
nanomole * hour/Liter (nmol*h/L) | 2.97 (128.00)

7. Secondary Outcome: Maximum Measured Concentration of 14C-BI 1467335-Equivalence (EQ) (Cmax) on Day 28 Following a qd Dosing of 10 mg BI 1467335 Tablet Over 40 Days With a Single Dose of 10 mg [14C]BI 1467335 on Day 28
Description: Maximum measured concentration of 14C-BI 1467335-Equivalence (EQ) (Cmax) on Day 28 following a qd dosing of 10 mg BI 1467335 tablet over 40 days with a single dose of 10 mg [14C]BI 1467335 on day 28 is presented.
Time Frame: PK samples were collected at 2 hours (h) prior dosing and at 646, 648:33, 648:75, 649, 650, 651, 652, 654, 656, 658, 660, 672, 684, 696, 720, 744, 768, 792, 816, 817, 864, 912, 936, 937, 960, 1008, 1181, 1349, 1517, 1685 and 1853 h after dosing on Day 1.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1467335 10 mg (MD)
Number analyzed (Participants) | 8
nanomole/Liter (nmol/L) | 347.0 (16.5)

8. Secondary Outcome: Area Under the Concentration-time Curve of 14C-BI 1467335-Equivalence (EQ) in Plasma Following a qd Dosing of 10 mg BI 1467335 Tablet Over 40 Days With a Single Dose of 10 mg [14C]BI 1467335 on Day 28
Description: Area under the concentration-time curve of 14C-BI 1467335-Equivalence (EQ) in plasma following a qd dosing of 10 mg BI 1467335 tablet over 40 days with a single dose of 10 mg [14C]BI 1467335 on day 28 is presented.
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole * hour/ Liter (nmol*h/L)
Arm/Group | BI 1467335 10 mg (MD)
Number analyzed (Participants) | 8
nanomole * hour/ Liter (nmol*h/L) | 67400.00 (7.58)

9. Secondary Outcome: Maximum Measured Concentration of BI 1467335 (Cmax) on Day 28 Following a qd Dosing of 10 mg BI 1467335 Tablet Over 40 Days With a Single Dose of 10 mg [14C]BI 1467335 on Day 28
Description: Maximum measured concentration of BI 1467335 (Cmax) on Day 28 following a qd dosing of 10 mg BI 1467335 tablet over 40 days with a single dose of 10 mg [14C]BI 1467335 on day 28 is presented.
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1467335 10 mg (MD)
Number analyzed (Participants) | 8
nanomole/Liter (nmol/L) | 69.6 (65.0)

10. Secondary Outcome: Area Under the Concentration Time-curve of BI 1467335 on Day 28 Over the Time Interval 24 h Following a qd Dosing of 10 mg BI 1467335 Tablet Over 40 Days With a Single Dose of 10 mg [14C]BI 1467335 on Day 28
Description: Area under the concentration time-curve of BI 1467335 on Day 28 over the time interval 24 h following a qd dosing of 10 mg BI 1467335 tablet over 40 days with a single dose of 10 mg [14C]BI 1467335 on day 28 is presented.
Time Frame: Pharmacokinetic samples were collected at 2 hours (h) prior to drug administration and at 646, 648:33, 648:75, 649, 650, 651, 652, 654, 656, 658, 660, 672 h after drug administration on Day 1.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole * hour/Liter (nmol *h/L)
Arm/Group | BI 1467335 10 mg (MD)
Number analyzed (Participants) | 8
nanomole * hour/Liter (nmol *h/L) | 268.00 (123.00)

ADVERSE EVENTS:
Time Frame: From first day of drug administration until end of the trial, up to 50 days for SD group and up to 78 days for MD group.
Description: Treated set (TS): This set included all participants who received at least 1 dose of trial medication.
Arm/Group | BI 1467335 10 mg (MD) | BI 1467335 10 Milligram (mg) (SD)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1467335 10 mg (MD) (N=8) | BI 1467335 10 Milligram (mg) (SD) (N=8)
Nasopharyngitis (Infections and infestations) | 6 | 2
Headache (Nervous system disorders) | 4 | 1
Somnolence (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Catheter site inflammation (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Feeling cold (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Medical device site reaction (General disorders) | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eye irritation (Eye disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT03382509/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT03382509/SAP_001.pdf